CLINICAL TRIAL: NCT01241331
Title: A Randomized, Controlled Evaluation of the Safety and Efficacy of a Topical Treatment for Moderate-Severe Facial Acne Vulgaris
Brief Title: BLI1100 for the Treatment of Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLI1100-201
Record Dates: First submitted 2010-11-11; First posted 2010-11-16 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Acne Vulgaris
Keywords: moderate to severe facial acne vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BLI1100 (Experimental): BLI1100 topical cream
  Interventions: Drug: BLI1100
- Vehicle cream (Placebo Comparator): Vehicle topical cream
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: BLI1100 — BLI110 topical cream
  Arms: BLI1100
Drug: Vehicle cream — Vehicle topical cream
  Arms: Vehicle cream

SUMMARY:
The purpose of this study is to compare the safety and efficacy of formulation BLI1100 to its vehicle in the treatment of moderate-severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Qualifying Investigator's Global Assessment severity score
* Qualifying number of non-inflammatory lesions
* Qualifying number of inflammatory lesions

Exclusion Criteria:

* Facial hair (beard), excessive scarring, sunburn or other disfigurement that may obscure the accurate assessment of acne grade
* Using medications that are reported to exacerbate acne
* Any clinically relevant finding at their baseline physical examination or dermatological medical history such as severe systemic diseases or diseases of the facial skin
* Have a known hypersensitivity or previous allergic reaction to any of the components
* Patients who have participated in an investigational clinical, surgical, drug, or device study within the past 30 days
* Patients who, in the opinion of the investigator, should not be included in the study for any reason, including inability to follow study procedures

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 233 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
percent reduction of total acne lesion counts | 12 weeks

SECONDARY OUTCOMES:
Investigator's Global Assessment | 12
  Rating of overall facial acne on a 4 point scale (0=clear to 4=severe) performed by a blinded investigator.
Change in serum chemistry | 12 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Center for Dermatology Clincal Research, Fremont, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists, Oceanside, California
  - Horizons Clinical Research Center, Denver, Colorado
  - North Florida Dermatology Associates, Jacksonville, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Atlanta Dermatology, Vein and Research Center, Alpharetta, Georgia
  - Peachtree Dermatology Associates Research Center, Atlanta, Georgia
  - Northwest Clinical Trials, Nampa, Idaho
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - The South Bend Clinic, South Bend, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Clinical Partners, Johnston, Rhode Island
  - DiscoveResearch, Bryan, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - The Education and Research Foundation, Lynchburg, Virginia
  - Virginia Clinical Research, Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington